CLINICAL TRIAL: NCT03888404
Title: Attitudes and Decision-making After Pregnancy Testing Study
Acronym: ADAPT
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-23592; R01HD108643 (NIH)
Record Dates: First submitted 2019-03-19; First posted 2019-03-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Unintended Pregnancy; Undesired Pregnancy
Keywords: Unintended Pregnancy; Unintended Birth; Pregnancy Preferences; Pregnancy Desires; Prenatal Care; Abortion; Adoption; Pregnancy Decision-Making; Mental Health; Stress; Socioeconomic Status; Education
MeSH Terms: conditions — Psychological Well-Being | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Underlying Cohort: The study will recruit and follow a prospective cohort of women "at risk" of pregnancy for one year.
  Interventions: Other: Pregnancy preferences (Aim 1)
- Pregnancy Match Cohort, Pregnant Group: Women from the Underlying Cohort who become pregnant will be transferred into the Pregnancy Match Cohort to be followed for two years.
  Interventions: Other: Sociocultural environment (Aim 2); Other: Pregnancy preferences (Aim 3a)
- Pregnancy Match Cohort, Not Pregnant Group: The study will also follow a comparison cohort of non-pregnant women from the Underlying Cohort, frequency matched to the pregnant participants on Desire to Avoid Pregnancy score and time at risk of pregnancy.
  Interventions: Other: Pregnancy (Aim 3b)

INTERVENTIONS:
Other: Pregnancy preferences (Aim 1) — The primary exposure of interest for Aim 1 will be pregnancy preferences, measured with the Desire to Avoid Pregnancy scale.
  Groups: Underlying Cohort
Other: Sociocultural environment (Aim 2) — For Aim 2 will assess the roles of contextual and individual variables on pregnancy decision-making and care-seeking outcomes (including state political environment, stigma, social emotional and instrumental support, feelings about the pregnancy, SES).
  Groups: Pregnancy Match Cohort, Pregnant Group
Other: Pregnancy preferences (Aim 3a) — The primary exposure of interest for Aim 3a will be pregnancy preferences, measured with the Desire to Avoid Pregnancy scale.
  Groups: Pregnancy Match Cohort, Pregnant Group
Other: Pregnancy (Aim 3b) — The exposure of interest for Aim 3b will be experiencing pregnancy. DAP level will be examined as an effect modifier.
  Groups: Pregnancy Match Cohort, Not Pregnant Group

SUMMARY:
The ADAPT Study is a longitudinal observational cohort study examining women's pregnancy preferences, pregnancy decision-making processes, and the effects of less preferred (commonly called "unintended") pregnancy on women's lives. This study will enroll and follow prospectively an Underlying Cohort (UC) of women who are not pregnant at baseline. The study will measure the degree to which participants desire to avoid pregnancy multiple times over the course of the year and capture incident pregnancies as they occur over time. Participants experiencing new pregnancies during the one-year UC will be transferred into a new cohort, the Pregnancy and Match Cohort (PMC); these women will be followed over the course of their pregnancy decision-making and health care-seeking to document these processes. In addition, they will be followed through their pregnancies and giving birth to investigate differences in health, well-being, and socioeconomic outcomes associated with carrying a pregnancy to term based on the participant's pre- and post-pregnancy preference about the pregnancy. Finally, a cohort of non-pregnant women from the UC, matched on desire to avoid pregnancy and time at risk of pregnancy, will be followed as part of the PMC. The study will compare the health, well-being, and socioeconomic outcomes of women with new pregnancies and new births to those in the non-pregnant group to assess the effect of pregnancy itself on women.

The ADAPT study has the following aims:

Aim 1: Assess the factors associated with women's pregnancy preferences, how preferences change over time, and their associations with contraceptive use, incident pregnancy, and feelings about the pregnancy after discovery (Underlying Cohort)

Aim 2: Investigate the options that women consider when they become pregnant and the factors that influence their pregnancy decision-making and ability to access desired reproductive health care and services (prenatal, abortion, adoption) (Study A)

Aim 3a: Examine the effects of giving birth from a less preferred (or "unintended") pregnancy, measured prospectively on a continuum, as compared to a more preferred pregnancy, on women's health and well-being (Study B1)

Aim 3b: Examine the effects of experiencing pregnancy and birth on women's health and well-being, as compared to not experiencing pregnancy (Study B2)

This is a social science, behavioral study and does not use clinical data or biological markers.

DETAILED DESCRIPTION:
The ADAPT Study is a longitudinal observational cohort study. The study has four components, each corresponding to a study aim: 1) Underlying Cohort (Aim 1); 2) Pregnancy and Match Cohort, Study A (Aim 2); 3) Pregnancy and Match Cohort, Study B1 (Aim 3a); and 4) Pregnancy and Match Cohort, Study B2 (Aim 3b).

This ADAPT study will recruit an "Underlying Cohort" (UC) of approximately 2,200 English or Spanish-speaking women, ages 15-34, who are not pregnant (or are terminating a pregnancy) and who are seeking care at designated primary and reproductive health care facilities in four states (see Eligibility Criteria). Participants will be followed up to a year as a part of the UC. At the UC baseline and follow-up surveys conducted every 6 weeks, participants will complete a psychometrically validated measure of prospective preferences and feelings about a potential pregnancy, the Desire to Avoid Pregnancy (DAP) scale. Analyses of UC data will examine the degree to which DAP scores change over time, as well as the relationships between DAP score and contraceptive use, pregnancy, feelings about incident pregnancies after they occur, collected at follow-up surveys.

Participants experiencing new pregnancies during the one-year UC will be transferred into a new cohort, the Pregnancy and Match Cohort (PMC), and will be followed for two years. In the PMC, participants will complete 8 surveys at: PMC baseline (right after reporting a new pregnancy), 6 weeks, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months. Surveys will capture the pregnancy options participants consider (raising child, abortion, adoption), health care and services participants seek (prenatal, abortion, adoption), services obtained and pregnancy outcome. Analyses will examine the factors influencing decision-making and ability to obtain desired care/services, including state sociopolitical environment around reproductive health.

PMC participants will also be a part of PMC-Study B1, in which they will be followed through the course of their pregnancies and childbirth to investigate health, well-being, and socioeconomic outcomes. All PMC surveys will include measures of stress and mental health; well-being; socioeconomics and employment; educational goals and attainment; alcohol, tobacco and drug use; physical health; and intimate partner violence so that individual trajectories of these outcomes will be available over time. Surveys administered after the birth of a child will also assess birth, maternal and child outcomes, including prematurity, low birth weight, breast-feeding, post-partum depression, maternal bonding, and child development. Study B1 will investigate how these outcomes differ based on the woman's prospective preference about the pregnancy, as well as her attitudes and feelings about it upon discovery. Analyses will compare outcomes among women giving birth by pregnancy preferences level; separately, analyses will also include the women who experienced miscarriage or terminated pregnancies. The hypothesis is that women with higher DAP scores will experience poorer outcomes after pregnancy and birth than those with higher DAP scores.

Finally, PMC-Study B2 will examine the effect of pregnancy itself on health and well-being outcomes. Throughout the UC as new pregnancies occur, a cohort, frequency matched on pregnancy preference score and time at risk of pregnancy, will also be followed as part of the PMC. Non-pregnant matches who experience pregnancy within a year of enrollment will themselves enter the pregnancy cohort and be assigned a non-pregnant match for the remainder of their time in the PMC. Analyses will compare the health, well-being, and socioeconomic outcomes of women with new pregnancies (and, separately, new births) to those the non-pregnant group to assess the effect of pregnancy itself on women. Analyses will account for the interaction between pregnancy preferences and pregnancy. The hypothesis is that experiencing a less preferred pregnancy (higher DAP score) will result in poorer health outcomes than avoiding a less preferred pregnancy.

Research activities will be conducted and coordinated by trained University of California, San Francisco (UCSF) research associates. Staff members at recruitment sites will not be engaged in the research. Data collection will involve completing confidential self-administered surveys using secure electronic systems (i.e., Qualtrics) or phone interviews over the course of the study. Participants will be followed for up to one year in the UC; those who transfer to the PMC will be followed for between 2-3 years overall. Participants will be remunerated with gift cards after each survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 to 34
* Is presenting for services at the participating recruitment site
* Speaks and reads English or Spanish
* Sexually active (has had sex in the last 3 months with a man/someone with sperm)
* Has a uterus (assigned female at birth)
* Resides in a study state or one directly bordering a study state
* Has access to a phone, internet, or smartphone
* Willing to be contacted by research team for 1-3 years by phone and either email or mail

Exclusion Criteria:

* Reports current pregnancy (unless having or initiating an abortion on the day of enrollment)
* Is sterilized or using an intrauterine device or transdermal implant at enrollment

Ages: 15 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female, trans-men, and gender non-conforming/queer people with uterus
Study Population: Women seeking care at participating reproductive health and primary care facilities
Sampling Method: Non-Probability Sample
Enrollment: 2015 (Actual)
Dates: Start 2019-03-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean score on Cohen's Perceived Stress Scale over 24 months (Aims 3a/3b) | PMC baseline through 24 months
  The Perceived Stress Scale (PSS) measures stress; scores are summed across 4 scale items (brief version), each with responses never to very often, on a 5-point scale, for a score ranging 0-16. The outcome will be the predicted mean PSS score over the 8 PMC survey observations (a single measure of effect), based on the marginal effect from a longitudinal multivariable mixed effects model.
Proportion experiencing moderate to severe depressive symptoms on the PHQ-8 over 24 months (Aims 3a/3b) | PMC baseline through 24 months
  Patient Health Questionnaire (PHQ-8) measures depression symptoms; scores are summed across the 8 items, each with responses not at all to nearly every day, on a 4-point scale, for a score ranging 0-24. Those scoring ≥ 10 are considered to have moderate to severe depression. The outcome will be the predicted probability of a PHQ-8 score ≥ 10 over the 8 PMC survey observations (a single measure of effect), based on the marginal effect from a longitudinal multivariable mixed effects model.
Proportion experiencing moderate to severe anxiety symptoms on the GAD-7 over 24 months (Aims 3a/3b) | PMC baseline through 24 months
  Generalized Anxiety Disorder (GAD-7) measures anxiety symptoms; scores are summed across the 7 items, each with responses not at all to nearly every day, on a 4-point scale, for a score ranging 0-21. Those scoring ≥ 10 are considered to have moderate to severe anxiety. The outcome will be the predicted probability of a GAD-7 score ≥ 10 over the 8 PMC survey observations (a single measure of effect), based on the marginal effect from a longitudinal multivariable mixed effects model.
Proportion of pregnancies ending in childbirth and childraising, among those who reported ever considering the option (Aim 2) | PMC baseline through 12 months
  Participants will report at each survey whether they considered each pregnancy option, as well as the status and outcome of their pregnancy. The outcome will be the proportion of participants whose pregnancies ended in childbirth and childraising, among those who ever reported considering giving birth and raising the child on a follow-up survey.
Proportion of pregnancies ending in abortion, among those who reported ever considering the option (Aim 2) | PMC baseline through 12 months
  Participants will report at each survey whether they considered each pregnancy option, as well as the status and outcome of their pregnancy. The outcome will be the proportion of participants whose pregnancies ended in abortion, among those who ever reported considering abortion on a follow-up survey.
Proportion of participants obtaining prenatal care, among those who ever reported seeking prenatal care (Aim 2) | PMC baseline through 12 months
  Participants will report at each survey whether they sought prenatal care, abortion care and/or adoption services and whether they obtained each type of care. The outcome will be the proportion of participants who obtained prenatal care, among those who ever reported seeking prenatal care.
Proportion of participants obtaining abortion care, among those who ever reported seeking abortion care (Aim 2) | PMC baseline through 12 months
  Participants will report at each survey whether they sought prenatal care, abortion care and/or adoption services and whether they obtained each type of care. The outcome will be the proportion of participants who obtained abortion care, among those who ever reported seeking abortion care.

SECONDARY OUTCOMES:
Proportion living below 100% of the Federal Poverty Level (FPL) (Aims 3a/3b) | PMC baseline through 24 months
  Participants will report on all surveys their household income and size. We will calculate the FPL cut-point based on the specific year's US Census Bureau FPL. The outcome will be the predicted probability of living below 100% FPL over the 8 PMC survey observations, based on the marginal effect from a longitudinal multivariable mixed effects model.
Mean MacArthur Scale of Subjective Social Status score over 24 months (Aims 3a/3b) | PMC baseline through 24 months
  Participants will rank themselves on the MacArthur Scale of Subjective Social Status (SSS) ladder (1-10) at all surveys. The outcome will be the predicted mean score over the 8 PMC survey observations, based on the marginal effect from a longitudinal multivariable mixed effects model.
Proportion employed full or part time (Aims 3a/3b) | PMC baseline through 24 months
  Participants will report on all surveys their current employment status. The outcome will be the predicted probability of being employed (full or part time) over the 8 PMC survey observations, based on the marginal effect from a longitudinal multivariable mixed effects model.
Time until dropping out of or leaving school (Aims 3a/3b) | PMC baseline through 24 months
  Participants will respond to questions at each survey about their current enrollment in school, type of school attended, degree sought, changes in enrollment since prior survey, degree completion/incompletion, and educational aspirations. Dropping out will be examined as, among those in a degree or other educational program at PMC baseline, time until stopping the degree for a reason other than completion.
Mean Diener's Flourishing Scale scores over 24 months (Aims 3a/3b) | PMC baseline through 24 months
  Diener's Flourishing Scale scores measures eudaimonic well-being; scores are summed across the 8 items, each with responses strongly agree to strongly disagree, on a 7-point scale, for total scores of 0-46. The outcome will be the predicted mean scale score over the 8 PMC survey observations, based on the marginal effect from a longitudinal multivariable mixed effects model.

OTHER OUTCOMES:
Proportion drinking any alcohol in the last month during pregnancy (Aims 3a/3b) | PMC baseline through 9 months, during pregnancy
  Participants will report at each survey how often they had a drink with alcohol in the last month. The outcome will be the predicted probability of drinking alcohol over PMC survey observations during which participants are pregnant, based on the marginal effect from a longitudinal multivariable mixed effects model.
Proportion drinking more than four drinks at a time in the last month (Aims 3a/3b) | PMC baseline through 24 months
  Participants will report at each survey how often they drank four or more alcoholic drinks at a time (heavy episodic drinking) in the last month. The outcome will be the predicted probability of heavy episodic drinking over the 8 PMC survey observations, based on the marginal effect from a longitudinal multivariable mixed effects model.
Proportion reporting physical and/or emotional intimate partner violence (IPV) from the man involved in the pregnancy in the last three months (Aim 3a) | PMC baseline through 24 months
  Participants will report at each survey whether the man involved in their pregnancy physically hurt them (physical IPV) or swore at or controlled their behavior (emotional IPV) in the last three months (minors excluded). The outcome will be the predicted probability of experiencing either type of IPV over the 8 PMC survey observations, based on the marginal effect from a longitudinal multivariable mixed effects model.
Proportion reporting their current physical health to be fair or poor, based on an adapted version of the SF-36 self-rated health item (Aims 3a/3b) | PMC baseline through 24 months
  Participants will respond at each survey to the question about how they rate their current physical health (excellent, very good, good, fair, poor). This self-rated health question is an adaptation of the item on the RAND Medical Outcomes Survey (SF-36) and the item used in the World Health Organization's World Health Survey. The outcome will be the predicted probability of fair/poor physical health over the 8 PMC survey observations, based on the marginal effect from a longitudinal multivariable mixed effects model.
Proportion of babies born prior to 37 weeks gestation (Aim 3a) | PMC follow-up survey (6 weeks through 24 months) at which birth is first reported
  In the PMC follow-up survey at which participants report having given birth, they will report the date that doctors expected the baby would be born and the actual birth date. Premature birth will be considered a birth occurring prior to three weeks before the due date.
Proportion at risk of poor bonding on the Postpartum Bonding Questionnaire (Aims 3a) | PMC follow-up surveys (6 weeks through 24 months), starting at the survey at which birth is first reported
  Participants will respond at each survey after the birth of the index child to the Brockington Postpartum Bonding Questionnaire, a 12-item scale, with responses on a 5-point scale from all of the time to never, total range 0-48. A score of ≥12 is considered to indicate risk of poor bonding. The outcome will be the predicted probability of being at risk of poor bonding over the 8 PMC survey observations, based on the marginal effect from a longitudinal multivariable mixed effects model.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Rocca, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rocca CH, Gould H, Gonzalez E, Foster DG, Munoz I, Parra M, Ralph LJ. Cohort profile: the ADAPT study, a prospective study of pregnancy preferences, pregnancy, and health and well-being in the southwestern USA. BMJ Open. 2024 Sep 25;14(9):e085372. doi: 10.1136/bmjopen-2024-085372. PMID 39322600